CLINICAL TRIAL: NCT04299633
Title: A Phase 1, Three-Part, Open-Label Study in Healthy Adult Subjects to Assess the Effect of Phosphate Binders on the Pharmacokinetics of a Single Dose of Vadadustat
Brief Title: Study in Healthy Adult Subjects to Assess the Effect of Phosphate Binders on the Pharmacokinetics of a Single Dose of Vadadustat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0037
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Pharmacokinetics; Phosphate binders; Sevelamer carbonate; Calcium acetate; Auryxia®; Vadadustat
MeSH Terms: interventions — vadadustat; Sevelamer; calcium acetate; ferric citrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: vadadustat plus sevelamer carbonate (Experimental): Participants will receive vadadustat 300 milligrams (mg) once on Days 1, 3, 5, and 7. Participants will receive sevelamer carbonate 1600 mg once on Days 3, 5, and 7.
  Interventions: Drug: Vadadustat; Drug: Sevelamer carbonate
- Part 2: vadadustat plus calcium acetate (Experimental): Participants will receive vadadustat 300 mg once on Days 1, 3, 5, and 7. Participants will receive calcium acetate 1334 mg once on Days 3, 5, and 7.
  Interventions: Drug: Vadadustat; Drug: Calcium acetate
- Part 3: vadadustat plus Auryxia® (Experimental): Participants will receive vadadustat 300 mg once on Days 1, 3, 5, and 7. Participants will receive Auryxia® 2 grams once on Days 3, 5, and 7.
  Interventions: Drug: Vadadustat; Drug: Auryxia®

INTERVENTIONS:
Drug: Vadadustat — 2 x 150 mg oral tablets
Drug: Sevelamer carbonate — 2 x 800 mg oral tablets
  Arms: Part 1: vadadustat plus sevelamer carbonate
Drug: Calcium acetate — 2 x 667 mg oral gelcaps
  Arms: Part 2: vadadustat plus calcium acetate
Drug: Auryxia® — 2 x 1 gram tablets (210 mg ferric iron equivalent to 1000 mg ferric citrate)
  Arms: Part 3: vadadustat plus Auryxia®

SUMMARY:
This 3-part study will be conducted to evaluate the interaction of vadadustat with sevelamer carbonate, calcium acetate, and Auryxia in healthy male and female participants. A total of 18 participants will be enrolled in each part of the study. Part 1 of the study will be conducted to assess the effect of a single oral dose of sevelamer carbonate (1600 milligrams [mg]) on the pharmacokinetics (PK) of a single oral dose of vadadustat (300 mg). Part 2 of the study will be conducted to assess the effect of a single oral dose of calcium acetate (1334 mg) on the PK of a single oral dose of vadadustat (300 mg). Part 3 of the study will be conducted to assess the effect of a single oral dose of Auryxia® (2 grams) on the PK of a single oral dose of vadadustat (300 mg).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age, inclusive, at time of informed consent

  1. Female participants of childbearing potential must be non-lactating, not pregnant as confirmed by a negative serum pregnancy test at screening and Day -1, and using, and agree to continue using, an effective method of contraception for at least of 4 weeks prior to the first dose of study drug until 30 days after the last dose of study drug. See the clinical trial protocol for acceptable methods of contraception prior to and during the study.
  2. Female participants of non-childbearing potential must be surgically sterile (e.g., hysterectomy, bilateral tubal ligation, oophorectomy) or post-menopausal (no menses for >1 year with follicle stimulating hormone [FSH] >40 Units per Liter (U/L) at screening).
  3. Female participants of childbearing potential must agree not to donate ova during the study and for at least 30 days after the last dose of study drug.
  4. Male participants who have not had a vasectomy for at least 6 months must agree to use an effective method of contraception during the study and until 90 days after the last dose of the study drug, and to not donate sperm during the study and for at least 90 days after the last dose of study drug. See the clinical trial protocol for acceptable methods of contraception prior to and during the study.
* Healthy per investigator judgment as documented by medical history, physical examination, vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and general observations

  1. At screening, abnormalities or deviations outside the normal ranges for any clinical assessments (laboratory tests, ECG, vital signs) may be repeated once at the discretion of the investigator(s), and results that continue to be outside the normal ranges must be judged by the investigator to be not clinically significant and acceptable for study participation.
  2. On Day -1, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin values must be within the upper limits of the normal range. All other laboratory test results that are outside the normal range on Day -1 and judged by the investigator to be not clinically significant may be repeated. Results that continue to be outside the normal range must be judged by the investigator to be not clinically significant and acceptable for study participation.
* Body mass index (BMI) between 18.0 and 30 kilograms per meters squared (kg/m^2), with a minimum body weight of 45 kg for females and 50 kg for males, inclusive
* Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure
* Willing and able to comply with the requirements of the study protocol

Exclusion Criteria:

* Current or past history of cardiovascular, cerebrovascular, respiratory, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease, as determined by the investigator. History of cancer (except treated non-melanoma skin cancer) or history of chemotherapy use within 5 years prior to screening.
* Any surgical or medical condition or history that, in the opinion of the investigator, may potentially alter the absorption, metabolism, or excretion of study treatment, such as, but not limited to gastric bypass surgery or gastric or duodenal ulcers
* Clinically significant history of dysphagia, bowel obstruction, or perforation
* Clinically significant history of hypercalcemia
* Clinically significant history of iron overload
* Clinically significant history of liver disease
* Clinically significant history of hypophosphatemia, ulcerative colitis, or gastrointestinal bleeding
* Contraindication to study drugs or its excipients and/or history of allergic or anaphylactic reactions
* Taking any of the following prohibited medications:

  1. Any prescription medication or over the counter multi-vitamin supplement, or any nonprescription products (including herbal-containing preparations but excluding acetaminophen up to 2 grams daily) within 14 days prior to Day -1;
  2. Any drug known to inhibit or induce cytochrome P450 (CYP) enzymes and/or P glycoprotein including St. John's wort (Hypericum perforatum) within 14 days or 5 half-lives (whichever is longer) prior to Day -1
* History of drug abuse within the previous year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening
* History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces [150 milliliters (mL)] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of screening or alcohol abuse within 1 year prior to screening
* Positive drug and alcohol test at screening or on Day -1
* History of latent or active tuberculosis (TB) as per documented medical history. Exposure to endemic areas within 8 weeks of screening
* Daily use of nicotine-containing products within 6 months of screening
* Consumed any food or drink/beverage containing grapefruit or grapefruit juice, apple or orange juice, pomelo juice, pomegranate, pineapple, star fruit, Seville or Moro (blood) orange products, and vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard) and charbroiled meats known to modulate CYP enzyme activity and transporters within 7 days before administration of study drug
* Positive test results of hepatitis B surface antigen (HBsAg), or positive hepatitis C virus antibody (HCVab) test result within 3 months prior to Day -1 or at screening
* Positive test results for human immunodeficiency virus (HIV) antibody within 3 months prior to Day -1 or at screening
* Participation in another clinical trial or exposure to any investigational agent within 30 days or 5 half-lives prior to Day -1, whichever is longer
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing
* Received a tattoo or body piercing (including ear piercings) within 2 months prior to Day 1, and/or open wound that may result in risk of infection
* Having a condition that the investigator believes would interfere with his/her ability to provide written informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the participant at undue risk
* Have previously participated in a clinical study that administered vadadustat

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Vadadustat area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, and 48 hours after each dose of vadadustat in each 9-day study part
Vadadustat area under the plasma concentration-time curve from time 0 to infinity (AUCinf) | 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, and 48 hours after each dose of vadadustat in each 9-day study part
Maximum observed plasma concentration (Cmax) of vadadustat | 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, and 48 hours after each dose of vadadustat in each 9-day study part

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Québec, Canada

IPD SHARING:
Plan to Share IPD: No